CLINICAL TRIAL: NCT02483403
Title: Longitudinal 3He Magnetic Resonance Imaging of Healthy Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: ROB0003
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Magnetic Resonance Imaging; Pulmonary Function; Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Other): Healthy elderly volunteers will undergo pulmonary function tests, hyperpolarized Helium-3 MRI at each visit.
  Interventions: Other: Hyperpolarized Helium-3; Device: MRI

INTERVENTIONS:
Other: Hyperpolarized Helium-3 — Hyperpolarized noble gas imaging using Helium-3 has been used to explore structural and functional relationships in the lung in patients with lung disease and healthy controls. In contrast to proton-based MRI imaging, Helium-3 gas is used as a contrast agent to directly visualize the airways, and thus ventilation. Whereas the normal density of gas is too low to produce an easily detectable signal, this is overcome by artificially increasing the amount of polarization per unit volume using optical pumping.
Device: MRI

SUMMARY:
Healthy elderly subjects male and female aged 65-85 will undergo MRI, lung function and exercise testing for the development of tools to quantify and validate longitudinal in vivo magnetic resonance imaging phenotypes of the aging lung.

DETAILED DESCRIPTION:
Briefly, during a single four hour visit, subjects will perform: 1) physical exam, 2) full pulmonary function tests, 3) cycle ergometry, 4) dyspnea and exertions scores using Borg scales, 5) BOLD Questionnaire and 6) 3He MRI before and after bronchodilation by deep inspiration, and potentially 25 minutes after inhalation of 2 puffs (200 µg) of the short-acting bronchodilator salbutamol in subjects who do not respond with 3He MRI ventilation improvements to deep inhalation. Hand-held spirometry will be performed post deep inspiration, and post salbutamol in those who receive salbutamol.

Subjects will first provide written informed consent and then be screened for MRI compatibility and will complete dyspnea and exertion scales, and full pulmonary function tests. A physical exam including vital signs and medical and smoking history will be performed. Subjects will complete the Bold Occupational Questionnaire and rest for approximately 15 minutes before cycle ergometry, including pre-and-post Borg scale evaluations. After completion of cycle ergometry, subjects will rest upright for 15 minutes and prepare for MRI which will be performed on 3 occasions within 1 hour: 1) before deep inspiration, 2) 3 minutes later after deep inspiration and, 3) 25 minutes later after inhalation of 2 puffs of salbutamol in subjects who do not respond to deep inhalation. Images obtained post deep inhalation will be assessed on the spot to determine if administration of salbutamol is required to resolve ventilation defects. Hand-held spirometry will also be performed post deep inspiration and post salbutamol in those who receive salbutamol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 60-90
* Subject has a smoking history of < 0.5 pack years
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject must be able to perform a breathhold for 16s.
* BMI 18-30
* Subject is judged to be in stable health on the basis of medical history
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)

Exclusion Criteria:

* Subject is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material.
* Subject has a history of cardiovascular disorders including coronary insufficiency, cardiac arrhythmias, severe hypertension (≥160 over ≥100)
* Subject has a daytime room air oxygen saturation <90% while lying supine.
* Subject is unable to perform spirometry or plethysmography maneuvers
* Subject is unable or unwilling to ride a stationary bicycle
* Subject is pregnant
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb,

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Ventilation Defect Percent (VDP) | 3 years
  Whole lung and segmental 3He MRI ventilation defect percent (VDP) are calculated by normalizing the volumes of 3He ventilation defects to the spatially matched CT whole lung and lung segments

SECONDARY OUTCOMES:
Apparent Diffusion Coefficients (ADC) | 3 years
  Diffusion weighted noble gas MRI provides a way to quantify pulmonary microstructure by sensing the movements of inhaled gas atoms. The "apparent" diffusion coefficient (ADC) during the diffusion time interval can be used to reflect the extent of alveolar restriction of gas atom movements, providing a surrogate measurement of airspace dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada